CLINICAL TRIAL: NCT02531672
Title: Detecting Recurrent Prostate Cancer With 11C-choline Positron Emission Tomography: An Expanded Access Study
Brief Title: Detecting Recurrent Prostate Cancer With 11C-choline Positron Emission Tomography
Status: No longer available | Type: Expanded Access
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-117
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer; Recurrent Prostate Cancer
Keywords: 11C-choline; Positron Emission Tomography; 15-117
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

INTERVENTIONS:
Drug: 11C-choline
Device: PET/CT Scan

SUMMARY:
The purpose of this study is to use a new imaging drug called 11C-choline that is used with a PET/CT scan to see prostate cancer when it cannot be seen well on other scans, such as bone scans, CT or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have biopsy-proven adenocarcinoma of the prostate initially treated with curative intent (surgery and radiation therapy are most common treatments but other treatments are also eligible).
* Biochemical recurrence defined as any of the following:

  1. PSA ≥ 0.2 ng/mL in at least two sequential tests for patients treated with surgery.
  2. PSA ≥ 0.2 ng/mL above the post therapy nadir for patients treated with radiation therapy, brachytherapy or cryotherapy.
  3. PSA ≥ 0.2 ng/ml above the most recent therapy nadir for patients who have received additional treatment in the recurrent setting
* Patient must have undergone standard-of-care restaging that does not clearly identify site(s) of active disease, or such prior studies must show equivocal findings for which further work-up is considered necessary to make clinical decision. Standard staging examinations may include one or more of the following: CT or MRI, bone imaging (either Tc-99m bisphosphonate scintigraphy MDP or F-18 sodium fluoride PET), FDG PET, or In-111 capromab pendetide scintigraphy no older than 3 months of consent date.
* Age ≥ 18 years.
* Patient must be able to tolerate PET/CT imaging.
* Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have claustrophobia that would preclude PET/CT imaging or other contraindications to CT imaging.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schӧder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/